CLINICAL TRIAL: NCT04101539
Title: A Randomized Trial Comparing Pulmonary Vein Isolation to Pulmonary Vein Isolation + OPTIMA Ablation in Patients Undergoing Ablation for Atrial Fibrillation
Brief Title: Comparing Pulmonary Vein Isolation to Pulmonary Vein Isolation + OPTIMA Ablation in Patients Undergoing Ablation for Atrial Fibrillation
Acronym: OPTIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00183327; U01HL141074 (NIH)
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation Chronic
Keywords: catheter ablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of patient and outcomes assessor to ablation protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Ablation (PVI) (Active Comparator): Patients in this arm will receive standard ablation for atrial fibrillation (wide-area circumferential ablation to achieve pulmonary vein isolation [PVI]).
  Interventions: Device: Standard PVI
- OPTIMA Ablation (Experimental): Patients in this arm will receive standard PVI ablation and supplemental ablation of reentrant driver sites identified by OPTIMA analysis as sites likely supportive of persistent atrial fibrillation.
  Interventions: Device: OPTIMA-guided catheter ablation

INTERVENTIONS:
Device: OPTIMA-guided catheter ablation — Patients in the experimental arm will undergo supplemental ablation of OPTIMA-identified sites hypothesized to support/perpetuate chronic atrial fibrillation.
  Arms: OPTIMA Ablation
Device: Standard PVI — Standard PVI for AF.
  Arms: Standard Ablation (PVI)

SUMMARY:
Catheter ablation is an established cornerstone of therapy for patients with symptomatic atrial fibrillation (AF) who wish to avoid anti-arrhythmic drug therapy or for whom anti-arrhythmics have proven ineffective. Pulmonary vein isolation (PVI), in which circumferential ablation is performed around the ostia of the pulmonary vein - left atrial junctions, is the standard ablation approach internationally. Single-procedure success rates (1y, freedom from AF, off anti-arrhythmics) for patients with paroxysmal AF is roughly 70%, and even worse (roughly 50%) for patients with persistent AF.

A number of strategies have been developed to improve outcomes in patients undergoing AF ablation, particularly in patients with persistent AF. Unfortunately, large prospective randomized trials (including STAR-AF II, published in NEJM in 2015) have demonstrated a failure of ancillary ablation techniques to improve AF ablation outcomes relative to PVI alone.

In a collaborative effort between the Cardiology electrophysiology group and the Trayanova laboratory (Biomechanical Engineering), investigators have developed a strategy of patient-specific modeling to identify pro-arrhythmic sites in AF patients that may be amenable to ablation. In this approach, patients undergo a pre-ablation cardiac MRI with late gadolinium enhancement, to delineate regions of healthy atrial tissue and regions of scar (this scan is clinically indicated, and performed currently in patients undergoing PVI for AF). A novel in silico modeling to determine regions supporting electrical reentry in the atrium, driving ongoing AF, has been developed by the Trayanova lab. In preliminary studies, investigators have demonstrated the ability to identify and target these regions with catheter ablation in patients undergoing PVI.

Investigators would like to conduct a prospective, randomized clinical trial in patients undergoing ablation for symptomatic persistent AF. All patients enrolled would undergo standard pre-procedure imaging (LGE-MRI) prior to the day of procedure. Investigators have developed methodology termed OPTIMA (OPtimal Target Identification via Modeling of Arrhythmogenesis) to determine, based on non-invasive patient-specific anatomic and tissue data from late gadolinium enhancement cardiac MRI (LGE-CMR) and simulation of cardiac electrical function, personalized ablation targets for persistent AF in patients with fibrotic remodeling.. Patients would be randomized to receiving PVI only versus PVI + OPTIMA ablation at the time of ablation. Patients would then be followed in standard clinical fashion at 3m, 6m, and 12m to assess for ablation efficacy and for procedural complications.

Investigators postulate a 20% improvement in freedom from AF with PVI + OPTIMA ablation form 50% to 70% (compared to PVI alone), investigators anticipate that in 1:1 randomization, a sample size of 80 patients in each arm will yield a power calculation of 80% with an alpha of 0.05. Investigators anticipate that enrollment and 1y clinical follow-up for 160 patients (total) undergoing AF ablation will require a 4y timeline.

DETAILED DESCRIPTION:
Background: Atrial fibrillation (AF) is the most commonly encountered clinical arrhythmia. Symptoms arising from AF are common, and may include palpitations, fatigue, exertional intolerance, and angina. Relief of symptoms is achieved by rhythm control strategies including drug therapy and catheter ablation for AF. Catheter ablation is more effective than drug therapy, is the preferred method of rhythm control for patients in whom drug therapy has been ineffective or intolerable, and is increasingly used as first-line therapy. However, success rates for AF control after catheter ablation are imperfect, with AF recurrence rates between 30 - 50% at 1 year. Currently, catheter ablation focuses almost exclusively on electrical isolation of the pulmonary vein (PV) ostia (PV isolation; PVI), to eliminate triggering activity from ectopic foci in the PVs that, in the vast majority of patients, initiate AF. A number of strategies have been developed to improve outcomes in patients undergoing AF ablation, particularly in patients with persistent AF. Unfortunately, large prospective randomized trials (including STAR-AF II, NEJM 2015) have demonstrated a failure of ancillary ablation techniques to improve AF ablation outcomes relative to PVI alone. The failure of PVI and ancillary ablation techniques to deliver reasonable outcomes is exacerbated in patients with persistent AF (PsAF), who develop fibrosis in the atria. These patients have AF ablation outcomes that are demonstrably worse than those seen in patients with persistent AF. Investigators have recently developed methodology (termed OPTIMA, OPtimal Target Identification via Modeling of Arrhythmogenesis) to determine, based on non-invasive patient-specific anatomic and tissue data from late gadolinium enhancement cardiac MRI (LGE-CMR) and simulation of cardiac electrical function, personalized ablation targets for persistent AF in patients with fibrotic remodeling. These targets, which are determined off line pre-procedure, are then used to steer patient treatment. This technology is intended to make the procedure accurate and efficacious in persistent AF patients with fibrosis, and to eliminate the need for repeat ablations, offering long-term freedom from AF.

Hypothesis: In patients undergoing ablation for the treatment of persistent AF, using the OPTIMA approach and performing PV isolation during ablation for AF will improve outcomes compared to performing PV isolation alone.

Importance: In United States, Center for disease control estimates that 2.7-6.1 million people suffer with AF and expects this number to increase with the aging population. Ablation for AF is performed at increasing rates, and in certain population (eg patients with paroxysmal AF) is moderately effective. Even in optimal patients, however, the rate of AF recurrence following apparently successful PV isolation is high (2017 Heart Rhythm Society (HRS) Consensus statement on AF ablation). Strategies to improve AF ablation outcomes should result in improved patient health (symptom elimination), lower patient risk (reduction of the number of patients undergoing redo ablation procedures), and reduced economic burden from healthcare costs (reducing post-ablation treatment for AF, including redo ablation procedures). Furthermore, demonstration of the arrhythmogenic propensity of fibrotic remodeling in patients with persistent AF will add to investigators' collective understanding of the fundamental mechanisms underlying AF initiation and perpetuation.

Objectives: The goal of this study is to test the efficacy of the OPTIMA approach for determining the optimal ablation targets in patients with persistent AF and fibrosis, and to demonstrate that elimination of AF-perpetuating sources in the fibrotic substrate, in conjunction with PVI, during AF ablation improves rate of AF-free survival at 1 year compared to patients undergoing standard PVI alone.

Study Procedures

This study is a prospective, randomized, single-blind study of patients undergoing either standard PV isolation or PVI+OPTIMA ablation for the treatment of symptomatic persistent AF. Patients referred for ablation for symptomatic persistent AF will be considered for enrollment. Patients will have cardiac function and anatomy assessed by echocardiography in the six-month window prior to ablation (routine care). Patients will have a baseline rhythm assessment with Ziopatch to quantify pre-ablation AF burden. All patients will undergo pre-procedure LGE-CMR to delineate atrial anatomy (routine care). MRI scan will be obtained in sinus rhythm; patients will be cardiovertered before MRI if the patients are in atrial fibrillation. All patients will be anticoagulated according to standard clinical guidelines. Patients with a CHADS VASc score of 2 or greater will be systemically anticoagulated in the pre-, peri-, and post-procedural periods. Patients not otherwise requiring long-term systemic anticoagulation will be anticoagulated during the peri- and post-procedural intervals (minimum of 2 months systemic anticoagulation following ablation). Finally, any patient undergoing cardioversion to facilitate MRI acquisition will receive systemic anticoagulation for a minimum of three weeks prior to cardioversion and/or have a Transesophageal Echocardiography (TEE) performed prior to cardioversion. After CMR acquisition, patients will be randomized to PVI versus PVI+OPTIMA ablation. Pre-procedural TEE is not required for patients presenting in Sinus rhythm and on uninterrupted anticoagulation for at least 3 weeks, regardless of CHADS VASC score. Patients presenting either in atrial fibrillation or not on uninterrupted anticoagulation will undergo a pre-procedural TEE, again independent of CHADS VASC score. All patients will undergo AF ablation with PVI (routine care). At the outset of the procedure, electroanatomical mapping of the Left Atrium (LA) will be performed to facilitate clinical ablation, with typically 1000 datapoints captured in the LA. PVI will be performed in all patients. In the PVI+OPTIMA arm, sites identified as targets by pre-procedure modeling will subsequently be targeted for ablation (research procedure, during routine ablation procedure). Additional ablation of other atrial targets (lines, complex fractionated electrograms) will be discouraged in both arms, but ultimately targeting such areas will be left to the discretion of the operator. In both arms, PV isolation will be assessed by entrance block. OPTIMA lesions will be assessed by both minimum of 50 percentage reduction in all local Electrograms (EGM), as well as non-capture by high output pacing at the site of target ablation. Operator will have the discretion not to ablate certain OPTIMA targets for safety reasons including but not limited to avoid critical structures and patient hemodynamic status. Operator will document the reason for not ablating all OPTIMA targets in the case report forms. Patients will be maintained on anti-arrhythmic drugs during the healing phase (3m) following ablation, with medication changes (cessation, up-titration, or drug changes) made at the discretion of the treating physician. All patients will be followed clinically after ablation in the standard fashion (routine care), including visits at 3, 6, and 12 months, with AF burden assessment with Zio patch at each visit.

Study duration and number of study visits required of research participants.

Investigators anticipate that this study will take 3 years for enrollment and 1 year clinical follow-up. Patient encounters include a pre-procedure clinical assessment and rhythm assessment(zio patch) in outpatient Electrophysiology (EP) Clinic; cardiac MRI in the week prior to ablation; the ablation procedure itself; overnight monitoring in the hospital following ablation; clinical assessment at 3, 6 and 12 months after ablation, including rhythm assessment with Ziopatch at each visit. Additional rhythm assessment with Ziopatch will be performed for patients with clinical symptoms of atrial fibrillation. Of note, these encounters are all part of current clinical practice in patients undergoing AF ablation.

Blinding, including justification for blinding or not blinding the trial, if applicable.

Patients will be blinded to the ablation strategy (PVI only versus PVI+OPTIMA ablation). Operators by necessity cannot be blinded to the ablation strategy, as patients are performing the ablations.

Risks

All patients in the study will undergo standard PVI, with its attendant risks. These risks include those related to general anesthesia, risk of stroke, risk of cardiac puncture, risk of esophageal injury, risk of other cardiac damage, and risk related to vascular access. Patients randomized to Re-entrant Driver (RD) ablation will undergo standard PVI (with risks listed above). During ablation, operators will target additional sites for lesion delivery. This is anticipated to lead to increases in procedure time, left atrial dwell time, number of lesions delivered, and increased radiation exposure.

Investigators anticipate that the additional risk to patients undergoing OPTIMA ablation (in addition to PVI) will be minimal. Typical PVI involves lesion delivery at 50-60 sites. In investigators early experience, patients have between 2-5 AF sources in the fibrotic substrate that OPTIMA targets. Thus, the additional ablation in each patient is likely to be a small component of the total ablation lesion set; additional risks are a function largely of time manipulating catheters and ablating in the left atrium. This added time will be minimal.

Radiation exposure Patients undergoing standard ablation procedure is estimated to be estimated to have 0.700 rems of radiation exposure due to fluoroscopy. Patients undergoing optima ablation are estimated to be exposed to additional 0.14 rems of radiation.

Risks of ECG patch monitor Clinical trials have so far shown the Zio XT is well-tolerated in the overall population. The risks associated with Zio patch include mild discomfort and/or allergic reaction to sticky pads used to attach the Zio patch.

There is a possibility that while reviewing one's patch monitor results investigators may detect a heart rhythm abnormality that investigators did not expect to find. Investigators will contact the patient and inform the patient and his/her clinical cardiac electrophysiologist regarding the result. The costs for any care that may arise in reaction to this incidental finding will not be covered by this research study.

Steps taken to minimize the risks.

Currently investigators employ a number of risk mitigation strategies, including the use of electroanatomical mapping systems to minimize radiation exposure, the use of systemic anticoagulation to minimize Cardiovascular Accident (CVA) risk, the use of ultrasound guided vascular access to minimize vascular complication rates. All of these strategies will be employed for all study participants. In addition following monitoring procedures will be followed during the study.

* Data quality will be monitored routinely and reviewed monthly for missing data, inconsistent data, data outliers, and potential protocol deviations.
* All adverse events and protocol deviations will be notified to PI.
* In order to minimize risks to patients enrolled in the study all adverse events will be discussed in the monthly cardiac electrophysiology complications conference. This conference will serve as the Global safety monitoring committee.
* All Attending physicians participating in this study including David Spragg MD, Ronal Berger MD, Hugh Calkins, MD, Joseph Marine, MD and Hiroshi Ashikaga MD, PhD attend this conference.
* All adverse events will be assessed in terms of relationship to device, relationship to procedure, severity, subsequent intervention required, and resolution status.

Benefits

Strategies to improve AF ablation outcomes should result in improved patient health (symptom elimination), lower patient risk (reduction of the number of patients undergoing redo ablation procedures), and reduced economic burden from healthcare costs (reducing post-ablation treatment for AF, including redo ablation procedures). Furthermore, demonstration of the importance of elimination of the arrhythmogenic propensity of the fibrotic substrate in patients with PsAF will add to investigators collective understanding of the fundamental mechanisms underlying AF initiation and perpetuation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must be at least 18 years old at the time of enrollment.
* Patient was referred to Johns Hopkins cardiac electrophysiology division for clinically indicated catheter ablation for persistent or long standing persistent AF either for index ablation or redo ablation.
* Patient is currently on systemic anticoagulation or has no contraindication to initiate systemic anticoagulation.
* Capable of undergoing informed consent.
* A Pre-Op cardiac MRI including LGE in sinus rhythm must be performed prior to ablation and patient should be capable of undergoing cardioversion and cardiac MRI.
* MRI scan should show evidence of left atrial scarring.

Exclusion Criteria:

* Patient is not a suitable candidate for AF ablation.
* Patient is currently not on anticoagulation and has significant contraindications to initiate systemic anticoagulation.
* Pregnant women may not participate in the study because gadolinium MRI contrast is contraindicated in pregnancy.
* Patient with Body weight more than 300 lbs as they cannot undergo MRI scans.
* Patients with Glomerular Filtration Rate (GFR) < 30 mL/min should not be enrolled in the study due to the use of intravenous gadolinium as an MRI contrast agent.
* No evidence of Left Arial fibrosis in MRI scan as these images are not suitable for simulation.
* Inability to get MRI in sinus rhythm.
* Long standing persistent AF more than 3 years of duration.
* Prior surgical maze procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmias (>30s) | 1 year
  Freedom from recurrent Atrial fibrillation (AF)/Atrial Tachycardia (AT)/Atrial Flutter (> 30s) after 90 day blanking period. This will be measured as the percentage of the study population that is free from atrial arrhythmias during the 1y follow-up period.

SECONDARY OUTCOMES:
Change in AF burden | 1 year
  This will measure the change in percentage time spent in AF for each study patient after ablation (baseline is the pre-ablation percentage time in AF). The change in AF burden for the overall study population will be calculated and expressed.
Percent participants with 70% or more reduction in AF burden | 1 year
  This will be a measure of the number of patients in each study group that achieve at least a 70% reduction in their baseline AF burden. This outcome will be expressed as a percentage of the number of patients in each study group meeting this outcome.
Freedom from major complications | 1 year
  This is a comparison of the percentage of patients in each study arm suffering a major complication. Complications including the following: death, stroke, cardiac tamponade, atrial-esophageal fistula, vascular injury, hemorrhage, cardiac injury, myocardial infarction, or other major complications resulting in either reparative procedure or prolonged hospitalization. Outcome will be expressed as a ratio.

CONTACTS AND LOCATIONS:
Overall Officials: David Spragg, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified patient data may be shared among study team members.